CLINICAL TRIAL: NCT02416219
Title: Efficacy of Surface Landmark Palpation for Identification of the Cricoid Cartilage in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Fatemah Qasem, Clinical fellow, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 106074
Record Dates: First submitted 2015-04-07; First posted 2015-04-14 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Aspiration Pneumonia
Keywords: Cricoid cartilage, cricoid pressure, obstetric
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cricoid Cartilage localization: The caregiver will be asked to palpate the cricoid cartilage and draw aline where he will apply cricoid pressure during rapid sequence induction
  Interventions: Procedure: Cricoid pressure; Device: Ultrasound

INTERVENTIONS:
Procedure: Cricoid pressure — participants will ask to mark the place where they will apply cricoid pressure if the patients was undergoing rapid sequence induction. US will be used to confirm how accurate they are in their estimation.
  Other Names: Sellick's Maneuver
Device: Ultrasound

SUMMARY:
Rapid Sequence Induction (RSI), with cricoid pressure is advocated for all obstetric patients undergoing general anesthesia. Applying cricoid pressure correctly is crucial to prevent aspiration. Using Ultrasound guidance we will be assessing the ability of different disciplines of caregivers to correctly localize the cricoid cartilage in obstetric patients by anatomical landmark palpation.

DETAILED DESCRIPTION:
Obstetric patients coming for elective cesarean delivery will be recruited for the study. Informed consent will be obtained from the patient. The participant (anesthesiologist, resident, nurse, or RT) will mark the center of the cricoid cartilage with the patient in the sniffing position, using fluorescent "invisible" ink. Another anesthesiologist who is expert in using ultrasound will find the proximal and distal margins of the cricoid cartilage an will draw a line at the middle of the 2 margins. Evaluation of the participant's assessment will be considered accurate if it falls within 5 mm from the ultrasound's measured line .The assessor will also be asked to score the ease of cricoid cartilage palpation between 1 to 10 using a visual analog scoring (VAS) scale. Total time taken for palpation will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years and older
* ASA 1-2•Having singleton pregnancy.
* Gestational age >37.
* Elective cesarean section

Exclusion Criteria:

* Patient refusal.
* Renal failure.
* Severe preeclampsia.
* Non- scheduled caesarean delivery (urgent).
* Twin pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Term Obstetric patients coming for elective cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Distance between measured Cricoid cartilage (by Assessors) and Ultrasound | 10 minutes
The level of difficulty to locate Cricoid cartilage NRS score | 10 minutes
Total time required for assessment | 10 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, MD, FRCPC, Principal Investigator — Western University, Schulish school of Medicine, Department of Anesthesia
Locations (1):
- London Health Science Centre, London, Ontario, Canada

REFERENCES:
- [Background] Zeidan AM, Salem MR, Mazoit JX, Abdullah MA, Ghattas T, Crystal GJ. The effectiveness of cricoid pressure for occluding the esophageal entrance in anesthetized and paralyzed patients: an experimental and observational glidescope study. Anesth Analg. 2014 Mar;118(3):580-6. doi: 10.1213/ANE.0000000000000068. PMID 24557105
- [Background] Benhamou D, Bouaziz H, Chassard D, Ducloy JC, Fuzier V, Laffon M, Mercier F, Raucoules M, Samii K. Anaesthetic practices for scheduled caesarean delivery: a 2005 French national survey. Eur J Anaesthesiol. 2009 Aug;26(8):694-700. doi: 10.1097/EJA.0b013e328329b071. PMID 19412111
- [Background] Fenton PM, Reynolds F. Life-saving or ineffective? An observational study of the use of cricoid pressure and maternal outcome in an African setting. Int J Obstet Anesth. 2009 Apr;18(2):106-10. doi: 10.1016/j.ijoa.2008.07.006. Epub 2009 Jan 13. PMID 19144507
- [Background] Aslani A, Ng SC, Hurley M, McCarthy KF, McNicholas M, McCaul CL. Accuracy of identification of the cricothyroid membrane in female subjects using palpation: an observational study. Anesth Analg. 2012 May;114(5):987-92. doi: 10.1213/ANE.0b013e31824970ba. Epub 2012 Feb 24. PMID 22366848
- [Background] Hung O, Scott J, Mullen T, Murphy M. Waiting to exhale! Anesth Analg. 2012 May;114(5):927-8. doi: 10.1213/ANE.0b013e31823a84ef. No abstract available. PMID 22523407
- [Background] Singh M, Chin KJ, Chan VW, Wong DT, Prasad GA, Yu E. Use of sonography for airway assessment: an observational study. J Ultrasound Med. 2010 Jan;29(1):79-85. doi: 10.7863/jum.2010.29.1.79. PMID 20040778